CLINICAL TRIAL: NCT07141927
Title: The Effects of Kinesiophobia and Proprioception on Disability and Function in Rheumatoid Hand
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Selvin BALKİ, associate professor, Ph.D., Cumhuriyet University
Other Study IDs: SCU-FTR-SB-03
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Disability; Function; Joint reposition sense; Kinesiophobia; Rheumatoid hand; Muscle strength
MeSH Terms: conditions — Arthritis, Rheumatoid; Kinesiophobia | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA group: RA volunteers followed in the rheumatology outpatient clinic of a university hospital
  Interventions: Other: Measurements
- Healthy controls: Hospital staff and volunteer companions of these RA patients
  Interventions: Other: Measurements

INTERVENTIONS:
Other: Measurements — First, the demographic characteristics of all participants were recorded. For those who met the inclusion criteria, primary and secondary outcome measurements were performed by the same physical therapist in a single session

SUMMARY:
This is a cross-sectional study aimed at examining the effects of kinesiophobia and proprioception on disability and function in the rheumatoid hand, compared to healthy controls.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a fairly common chronic inflammatory disease. Up to 90% of wrist and finger joints are affected by RA. Thus, it is known that a decrease in performance-based function and disability occur in the hand. Kinesiophobia leads to avoidance behavior, especially in painful conditions. Kinesiophobia has been shown to be a significant mental factor leading to functional loss and disability in rheumatoid hand (RH). On the other hand, joint repositioning sense measurements, which show proprioceptive losses in the wrist and hand joints due to the effects of RA, have been demonstrated. However, as far as we know, the contributions of these mental and biological factors (kinesiophobia + proprioception) to the function and disability of RH have not been examined together.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with RA

* Diagnosis of RA
* Volunteering
* Being between the ages of 18 and 65

Inclusion criteria for healthy controls

* Being healthy.
* Being between 18-65 years old.
* Being a volunteer

Exclusion Criteria:

Exclusion criteria for patients with RA:

* The presence of another rheumatic disease or chronic illness that could affect function and cause disability.
* Pain, deformity, or other cooperation issues (such as severe mental, visual, or hearing impairments) that prevent participation in measurements.
* Sensory loss in the upper extremity, history of surgery, and injury in the last six months.

Exclusion criteria for healthy controls

* Any diagnosis of chronic or acute illness.
* In the upper extremity, history of surgery injury in the last six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer patients receiving treatment and follow-up at the rheumatology outpatient clinic of a university hospital formed the study sample.
  The healthy control group included hospital staff and volunteer companions of these patients.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia | First day
  The participant's fear-avoidance behavior toward physical activity was assessed using the Tampa Kinesiophobia Scale.
Wrist-thumb proprioception | First day
  Joint position sense for wrist extension and thumb carpometacarpal flexion was assessed with goniometry. Joint position sense was measured by the ability to actively replicate a pre-determined target angle (30 degrees). During the measurement, the participant's evaluated joints was brought to the target angle and held in this position for three seconds. The participant was asked to hold this position in their memory, after which the joints will be passively returned to the starting position. Then, the participant was asked to actively move their hand to these pre-determined positions. The result was determined by the average deviation angle obtained from the measurements repeated at thirty-second intervals. These measurement were only taken with the dominant hand.
Hand function | First day
  Hand function was evaluated with the Dellon Modifiye Moberg pickup test.
Hand disability | First day
  Hand disability was evaluated with the Disabilities of the Arm, Shoulder, and Hand

SECONDARY OUTCOMES:
Demographic characteristics | First day
  Gender, age, employment and income status, smoking habits, and dominant hand information were recorded. Education below high school was categorized as low education. RA patients were also asked about the duration of their illness.
Disease activity | First day
  RA disease activity was assessed using the DAS28- theDiseaseActivity Score 28
Physical activity level | First day
  : Participants' physical activity levels were assessed using the International Physical Activity Questionnaire-Short Form. An IPAQ score of less than 600 metabolic equivalents (METs) was defined as low activity
Isometric wrist extensor muscle strength measurement | First day
  Measurements were taken with the participant sitting upright, elbow close to the body and bent at 90 degrees, forearm supported on a surface in pronation, and the wrist-hand in space. Strength measurement was performed using the MAKE method with the wrist in 30 degrees of extension and a dynamometer placed on the back of the hand.. The average of three measurements taken one minute apart after a trial was recorded in kilograms. This measurement was only taken with the dominant hand.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No